CLINICAL TRIAL: NCT07164105
Title: Mechanisms of Low Intensity Focused Ultrasound of the Ventral Anterior Cingulate Cortex for Post-Traumatic Stress Disorder in Frontline Healthcare Workers
Brief Title: LIFU Mechanisms for PTSD in Healthcare Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20252812
Record Dates: First submitted 2025-08-22; First posted 2025-09-09 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: PTSD and Trauma-related Symptoms
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low intensity focused ultrasound (LIFU) (Experimental): LIFU of the ventral anterior cingulate cortex
  Interventions: Device: Low intensity focused ultrasound
- Sham (Sham Comparator): Sham neuromodulation (Sorbothane membrane over ultrasound probe)
  Interventions: Device: Sham modulation

INTERVENTIONS:
Device: Low intensity focused ultrasound — Low intensity focused ultrasound neuromodulation of the ventral anterior cingulate cortex
  Other Names: LIFU
  Arms: Low intensity focused ultrasound (LIFU)
Device: Sham modulation — Low intensity focused ultrasound with a Sorbothane membrane cover to prevent acoustic energy transmission
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to evaluate whether low-intensity focused ultrasound (LIFU) of the ventral anterior cingulate cortex (vACC) can normalize dysfunctional brain activation patterns and behaviors in frontline healthcare workers with post-traumatic stress disorder. The main questions it aims to answer are:

* Does LIFU of the vACC effect activity and connectivity of the vACC and amygdala?
* Does LIFU of the vACC reduce post-traumatic stress symptoms? Researchers will compare LIFU to sham modulation to see if LIFU modulates activity of vACC-amygdala circuitry and affects threat sensitivity and emotion regulation.

Participants will:

* Complete two fMRI sessions (before and after LIFU)
* Receive a single session of LIFU or sham modulation of the vACC
* Wear a wearable device that tracks sleep and heart rate metrics

ELIGIBILITY:
Inclusion Criteria:

1. Adults in a frontline healthcare position (e.g. emergency medical services)
2. Ages 18-65 years
3. PTSD Checklist for DSM-5 (PCL-5) score ≥ 33 and < 65
4. English proficiency as evaluated by language ability during screening

Exclusion Criteria:

1. Neurological disorders
2. DSM-5 diagnosis of psychotic disorders, eating disorder, obsessive-compulsive disorder, moderate to severe alcohol or substance use disorder within the past year, bipolar disorder, or major depressive disorder with psychosis
3. Suicidal intent or plan (as measured by Suicide-Risk-Assessment-C-SSRS "Yes" answers to items 3, 4 or 5 of Suicidal Ideation-Past 1 month section, or any "Yes" answer to any of the items of Suicidal Behavior-Past 3 months section), or any suicide attempt in the last 3 months.
4. History of severe traumatic brain injury (as indicated by score ≥ 3 on the Tulsa Head Injury Screen) or of skull fractures
5. Contraindications to MRI as determined by the MR Environment Screening
6. Pregnancy, determined by urine pregnancy test administered prior to every MRI scanning procedure
7. Evidence of inability to comply with study procedures based on experimenter judgement.
8. Change in the dose or prescription of a medication within the 6 weeks before enrolling in the study that could affect brain functioning, e.g., anxiolytics, antipsychotics, antidepressants, benzodiazepines, or mood stabilizers.
9. Non-correctable vision or hearing problems
10. Unstable medical diagnoses
11. Any structural abnormalities in the LIFU target region on screening brain MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-29 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
LIFU target engagement | Study day 1 to day 7 (plus or minus 3 days)
  Percent BOLD signal change in vACC and amygdala regions of interest
Behavioral changes | Day 0 to Day 7 (plus or minus 3 days)
  Change in reaction time (ms) and error rate (percentage of correct answers) on emotional conflict task; difference between optimal and observed flight initiation distance.

SECONDARY OUTCOMES:
LIFU effects on physiology | Day 0 to day 14 (plus or minus 6 days)
  Change in heart rate variability (ms), change in resting heart rate (beats per minute), change in %REM sleep (minutes), change in %deep sleep (minutes) as measured by WHOOP® band
LIFU effects on PTSD symptoms | Dy 0 to day 14 (plus or minus 6)
  Change in PCL-5 score
fMRI-heart rate variability correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and heart rate variability (ms) as measured by WHOOP® band.
fMRI-resting heart rate correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and resting heart rate (beats per minute) as measured by WHOOP® band.
fMRI-REM sleep correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and %REM sleep (minutes) as measured by WHOOP® band.
fMRI-deep sleep correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and %deep sleep (minutes) as measured by WHOOP® band
fMRI-PTSD Symptom Correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and PCL-5 score.
fMRI-Emotion Regulation Correlation | Day 0 to day 14 (plus or minus 6)
  Correlations between vACC/amygdala BOLD signal extracted beta-weights and Cognitive-Emotion Regulation Questionnaire Score.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States